CLINICAL TRIAL: NCT06188169
Title: Effectiveness of Ultrasound-guided Lung Ventilation in Determining the Optimum Inspiratory Pressure in Pediatric Patients Undergoing Abdomino-pelvic Surgeries ; a Randomized Controlled Study
Brief Title: Effectiveness of Ultrasound-guided Lung Ventilation in Determining the Optimum Inspiratory Pressure in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Yahia El Sayed Kamel, Lecturer of anesthesiology and surgical ICU and pain management, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: US-guided Lung ventilation
Record Dates: First submitted 2023-10-29; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Pediatric Lung Atelectasis

STUDY DESIGN:
Intervention Model Description: This is a comparative prospective randomized controlled study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will be randomly allocated by a computer-generated list into one of the study groups. The randomization sequence will be concealed in sealed envelopes and will be opened by an independent nurse.
  Patients and data collectors will be blind to group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A = C-PCV received conventional pressure-controlled ventilation (Experimental): Inspiratory pressure will be adjusted to achieve an expired tidal volume of 7 ml/Kg; the respiratory rate will be adjusted to achieve an end ETCO2 at 32-35 mmHg, inspiratory to expiratory ratio at 1:2, PEEP at 4 cm H2O, and FiO2 at 0.5. No further adjustment in IP will be made throughout the surgery. LUS will be performed at the same fixed four-time interval as Group-B. Anesthesiologist will not do any interventions to the atelectatic areas in this group.
  Interventions: Procedure: Increasing the inspiratory pressure if atelectasis detected by US
- Group B = US-PCV: received ultrasound-guided pressure-controlled ventilation (Active Comparator): Initial IP will be ten cmH2O, PEEP 4 cmH2O with a 0.5 inspired oxygen fraction, and RR 12 breaths/min. Then under ultrasound guidance, a stepwise increase in inspiratory pressure from 10 cmH2O by 2 cmH2O increments every 5 min until the atelectasis disappeared on ultrasound (progression from lung collapse to B lines to normal lung image). The IP will be fixed at this level, and RR will be adjusted to maintain an EtCO2 at 32-35 mmHg. The maximum airway pressure will be limited to 35 cmH2O.
  Interventions: Procedure: Increasing the inspiratory pressure if atelectasis detected by US

INTERVENTIONS:
Procedure: Increasing the inspiratory pressure if atelectasis detected by US — The study used US to detect presence of lung atelectasis under mechanical ventilation in pediatrics. Inspiratory pressure increased gradually with continuous monitoring by lung US to minimize the atelectasis as possible.

SUMMARY:
This study aimed to show the Effectiveness of Ultrasound-guided Lung Ventilation to determine the appropriate level of inspiratory pressure sufficient to provide adequate pulmonary ventilation with the resolution of the atelectatic lung.

DETAILED DESCRIPTION:
Respiratory physiology is different in young children, especially in neonates and infants, from that of older children and adults. Neonates and infants have immature respiratory control, weak respiratory muscles, different airways, lung mechanics and higher basal metabolic oxygen requirements. Appreciating these distinctive respiratory characteristics in young children is necessary to formulate suitable anesthetic plans for the safe conduct of anesthesia as respiratory-related morbidity and mortality occur even in healthy children.

Atelectasis is a side effect of general anesthesia which can be found in all types of interventions and patients of all ages. The reported incidence of anesthesia-induced atelectasis in children varies from 12 to 42% in sedated and non-intubated patients and from 68 to 100% in children with general anesthesia with tracheal intubation or laryngeal mask.

Such lung collapse causes arterial blood oxygenation to decline during and after anesthesia. Although anesthesia-induced atelectasis resolves spontaneously in children with American Society of Anesthesiology's (ASA) physical status classification I to II after minor surgical procedures, this entity may persist in the postoperative period in high-risk children undergoing complex surgeries. In the latter population, atelectasis potentially increases the risk for ventilator-induced lung injury and could be associated with postoperative pulmonary complications.

Atelectasis and poorly ventilated lung areas appear during general anesthesia in adults as well as in children. It is of concern that collapsed lung tissue reduces lung compliance and causes venous admixture and arterial oxygenation impairment. Despite its high prevalence during anesthesia, bedside diagnosis of atelectasis remains challenging. Anesthesia-induced atelectasis is commonly small and thus mostly invisible on standard chest radiographs. In contrast, it can easily be diagnosed by tomographic imaging techniques such as computed tomography or magnetic resonance imaging (MRI). However, these latter are clinically impractical, expensive, time-consuming, and with harmful exposition to x-ray.

Sonography is a simple, non-invasive, and radiation-free methodology that has increased daily practice usage. Lung sonography (LUS) plays an important role in diagnosing pulmonary diseases in children, including obstructive and compressive atelectasis of different origins. Just as in adults, LUS could identify children needing a recruitment maneuver to re-expand their lungs and help optimize ventilator treatment during anesthesia. LUS could also identify critically ill children with a high risk for developing pulmonary complications due to residual atelectasis after surgery.

A prospective, randomized, double-blind study in the Second Affiliated Hospital and Yuying Children Hospital of Wenzhou Medical University showed that an inspiratory pressure of 12 cm H2O was sufficient to provide adequate ventilation with a lower occurrence of gastric insufflation during induction of general anesthesia in paralyzed Chinese children aged from 2 to 4 years old.

Many studies used LUS to determine the optimum positive end-expiratory pressure (PEEP), yet no previous studies used LUS to determine the best inspiratory pressure (IP) for pressure controlled ventilation. So, this study aimed to determine the appropriate level of inspiratory pressure sufficient to provide adequate pulmonary ventilation with the resolution of anesthesia-induced lung atelectasis using real-time ultrasonography in paralyzed children.

ELIGIBILITY:
Inclusion Criteria:

* Children's age starting from 5 to 12 years.
* Genders eligible for the study: both sexes.
* ASA I-II.
* They were scheduled for elective Abdomino-pelvic surgery lasting > 1.5 hours duration.

Exclusion Criteria:

* Parent refusal
* Emergency cases
* Laparoscopic surgeries
* Acute respiratory disease, pulmonary or lung diseases
* Lung consolidation score ≥ 2 before intubation
* Morbid obesity

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-08-12 (Actual)

PRIMARY OUTCOMES:
Incidence of significant anesthesia-induced lung collapse diagnosed by LUS examined at T2. | 1 minute after skin closure and before extubation (T2)
  Significant lung atelectasis will be defined as any region that had a lung consolidation score of ≥2.

SECONDARY OUTCOMES:
Time in minutes to resumption of normal lung aeration in the consolidated area started from diagnosis of collapse (T1) until lung consolidation score < 2 in group US-PCV | "from diagnosis of collapse until lung consolidation score < 2 in group US-PCV (assessed up to 5 minutes)"
Incidence of lung collapse in the two groups as detected by lung US at the 3rd formal lung ultrasound examination (T2). | 1 minute after skin closure and before extubation

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Soaida, MD, Study Director — Cairo University; Hany Mohammed, MD, Study Director — Cairo University; Mohamed Mohamed, MD, Study Director — Cairo University; Omnia Kamel, MD, Study Director — Cairo University
Locations (1):
- Abul Rish Pediatric Hospital, Giza, الجيزة, Egypt

IPD SHARING:
Plan to Share IPD: No